CLINICAL TRIAL: NCT02271412
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple Ascending Dose Study in Healthy Subjects to Evaluate the Safety, Tolerability, and Pharmacokinetics of LY03005
Brief Title: Multiple Ascending Dose Study in Healthy Subjects to Evaluate the Safety, Tolerability, and Pharmacokinetics of LY03005
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: LY03005 MAD; LY03005/CT-USA-102 (Other: Luye)
Record Dates: First submitted 2014-10-20; First posted 2014-10-22 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Major Depressive Disorder, Recurrent, Unspecified
MeSH Terms: conditions — Depressive Disorder, Major; Recurrence

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LY03005 (Experimental): LY03005 40, 80, 120, or 160 mg
  Interventions: Drug: LY03005
- Placebo (Placebo Comparator): Placebo at 40, 80, 120, or 160 mg
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY03005 — LY03005 is a new investigational pro-drug of desvenlafaxine formulated as extended-release oral tablets for the treatment of major depressive disorder.
  Other Names: 4-Methylbenzoate of desvenlafaxine hydrochloride
  Arms: LY03005
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Objectives

* To evaluate the safety and tolerability of escalating multiple oral doses of LY03005 in healthy subjects.
* To characterize the pharmacokinetics of escalating multiple oral doses of LY03005.

DETAILED DESCRIPTION:
This will be a randomized, double-blind, placebo-controlled, multiple ascending dose study to be conducted in the US. Approximately 48 healthy subjects will be enrolled into one of the four groups

ELIGIBILITY:
Inclusion Criteria:

1. Are capable of giving informed consent and complying with study procedures;
2. Are between the ages of 18 and 45 years, inclusive;
3. A negative pregnancy test result prior to screening and admission for all female subjects, and meet the following criteria defined as:

   1. If child-bearing potential, agree to avoid pregnancy during the study and one month after the end of the study by using effective contraceptive method(s), such as an intrauterine device (IUD), diaphragm with spermicide, and condoms with spermicide.
   2. Surgically sterile for at least 3 months prior to screening
   3. Postmenopausal
4. Considered healthy by the Principal Investigator, based on a detailed medical history, full physical examination, clinical laboratory tests, 12-lead ECG and vital signs;
5. Nonsmoker, defined as not having smoked or used any form of tobacco in more than 6 months before screening;
6. Body mass index (BMI) of 19 to 30 kg/m2 inclusive and body weight not less than 50 kg;
7. Willing and able to adhere to study restrictions and to be confined at the clinical research center.

Exclusion Criteria:

Subjects will be excluded from study entry if any of the following exclusion criteria are present at screening or admission:

1. Clinically significant history of gastrointestinal, cardiovascular, musculoskeletal, endocrine, hematologic, psychiatric, renal, hepatic, bronchopulmonary, neurologic, immunologic, lipid metabolism disorders, or drug hypersensitivity;
2. Subjects with a mean systolic blood pressure of three measurements less than 130 mmHG, or a mean diastolic blood pressure of three measurements less than 90 mmHG at screening. Blood pressure will be measured at supine position.
3. Known or suspected malignancy;
4. Positive blood screen for human immunodeficiency virus (HIV), or hepatitis B surface antigen (HBsAg), or hepatitis C virus;
5. A history of seizure. However, a history of febrile seizure is allowed;
6. Positive pregnancy test result, or plan to become pregnant if female;
7. A hospital admission or major surgery within 30 days prior to screening;
8. Participation in any other investigational drug trial within 30 days prior to screening;
9. DSM-V substance use disorder within 6 months prior to screening;
10. A positive result for alcohol or drugs of abuse at screening or admission;
11. Tobacco use within 6 months prior to screening;
12. An unwillingness or inability to comply with food and beverage restrictions during study participation;
13. Donation or blood collection of more than 1 unit (approximate 450 mL) of blood (or blood products) or acute loss of blood during the 90 days prior to screening;
14. Use of prescription or over-the-counter (OTC) medications, and herbal medicines (including St John's Wort, herbal teas, garlic extracts)within 14 days prior to dosing (Note: Use of acetaminophen at < 3g/day is permitted until 24 hours prior to dosing);
15. A history of intolerance or hypersensitivity to venlafaxine or desvenlafaxine or any excipients;
16. A history of suicide attempt in the past 12 months and/or seen by the investigator as having a significant history of risk of suicide or homicide; 17 An unwillingness of male participants to use appropriate contraceptive measures if engaging in sex intercourse with a female partner of childbearing potential. Appropriate measures include use of a condom and spermicide and, for female partners, use of an intrauterine device (IUD), diaphragm with spermicide, oral contraceptives, injectable progesterone, progesterone sub-dermal implants, or a tubal ligation. Sexual intercourse with pregnant or lactating women is prohibited.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2014-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events | 3 to 4 months
  Safety and Tolerability of LY03005

CONTACTS AND LOCATIONS:
Overall Officials: David Krefetz, MD, Principal Investigator — PRA - CRI Lifetree
Locations (1):
- PRA Health Sciences, Marlton, New Jersey, United States